CLINICAL TRIAL: NCT05941897
Title: A Phase II, Open-label, Multicentre, Non-comparative, Single-arm Local Study of Ceralasertib Plus Durvalumab in Patients With Advanced or Metastatic Non-Small Cell Lung Cancer Without Actionable Genomic Alterations, and Whose Disease Has Progressed On or After Prior Anti-PD-(L)1 Therapy and Platinum-based Chemotherapy
Brief Title: A Study to Investigate Efficacy and Safety of Ceralasertib Plus Durvalumab in Participants Aged ≥ 18 Years With Advanced or Metastatic Non-small Cell Lung Cancer Whose Disease Progressed on or After Prior Anti-PD-(L)1 Therapy and Platinum-based Chemotherapy
Acronym: LOTOS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZ-RU-00001
Record Dates: First submitted 2023-06-12; First posted 2023-07-12 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Advanced or Metastatic NSCLC
Keywords: Lung Neoplasms; Lung Diseases; Carcinoma, Non-Small-Cell Lung; Carcinoma, Bronchogenic; Respiratory Tract Diseases; Bronchial Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Durvalumab; Ceralasertib; ATR inhibitor; Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Lung Diseases; Carcinoma, Bronchogenic; Respiratory Tract Diseases; Bronchial Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms | interventions — ceralasertib; durvalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group A (Experimental): Ceralasertib plus durvalumab combination therapy Participants will be administered orally ceralasertib followed by IV durvalumab each 28 days cycle.
  Interventions: Drug: Ceralasertib; Drug: Durvalumab

INTERVENTIONS:
Drug: Ceralasertib — Participants will receive ceralasertib oral tablets.
Drug: Durvalumab — Participants will receive durvalumab as an intravenous infusion

SUMMARY:
A study to investigate efficacy and safety of ceralasertib plus durvalumab in participants aged ≥ 18 years with advanced or metastatic non-small cell lung cancer whose disease progressed on or after prior anti-PD-(L)1 therapy and platinum-based chemotherapy.

DETAILED DESCRIPTION:
This is a single-arm study, all participants will be assigned to one treatment group - ceralasertib plus durvalumab combination therapy. Each 28-day cycle will begin with ceralasertib administered orally followed by durvalumab administered intravenously.

The objectives of the current single-arm local study are to estimate the efficacy and safety of ceralasertib and durvalumab combination in local population to obtain relevant information for routine clinical practice. The results of this additional study will provide clinical data on efficacy and safety of an innovation drug in the new region - Russian Federation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented NSCLC that is locally advanced or metastatic according to Version 8 of the IASLC Staging Manual in Thoracic Oncology.
* Documented epidermal growth receptor factor (EGFR) and anaplastic lymphoma kinase (ALK) wild-type status.
* Documented radiological PD whilst on or after receiving the most recent treatment regimen.
* Eligible for second- or third-line therapy and must have received an anti-PD-(L)1 therapy and a platinum doublet containing therapy for locally advanced or metastatic NSCLC.
* Eastern Cooperative Oncology Group (ECOG)/World Health Organization (WHO) performance status of 0 or 1.
* Adequate organ function and marrow reserve.
* Body weight > 30 kg and no cancer-associated cachexia.

Exclusion Criteria:

* Participant with mixed SCLC and NSCLC histology.
* Brain metastases or spinal cord compression unless the participant is stable and off steroids.
* Persistent toxicities (CTCAE Grade > 2) caused by previous anticancer therapy.
* Active or prior documented autoimmune or inflammatory disorders.
* History of leptomeningeal carcinomatosis.
* Participants who have received more than one line of prior anti-PD-(L)1.
* Participants must not have experienced a toxicity that led to discontinuation of the prior anti-PD(L)1 therapy.
* Participants must not have experienced a Grade ≥ 3 immune-mediated adverse event (imAE) or an immune-related neurologic or ocular AE of any grade while receiving prior anti-PD(L)1 therapy.
* Participants must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged.
* Participants who have received more than one prior line of platinum-based chemotherapy in metastatic setting.
* As judged by the investigator, any evidence of medical condition, which, in the investigator's opinion, makes it undesirable for the participant to participate in the study.
* Participants who have received a prior ATR inhibitor.
* Diagnosis of ataxia telangiectasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | At month 6 after the last patient's first dose (approximately 18 months).
  Objective response rate (ORR) is defined as the proportion of participants who have a complete response (CR) or partial response (PR) per RECIST 1.1.

SECONDARY OUTCOMES:
Duration of Response (DoR) | Up to 30 months
  DoR is defined as the time from the date of first documented response until date of documented progression per RECIST 1.1.
Time to response (TTR) | Up to 30 months
  Time to response (TTR) is defined as the time from the start of treatment until the date of first documented objective response per RECIST 1.1.
Disease control rate (DCR) | At month 6 after the last patient's first dose (approximately 18 months).
  DCR at 18 weeks is defined as the percentage of participants who have a CR or PR or who have stable disease (SD) for at least 17 weeks per RECIST 1.1.
Progression free survival (PFS) | Up to 30 months
  PFS is defined as time from the start of treatment until progression per Response Evaluation Criteria in Solid Tumours, Version 1.1 (RECIST 1.1).
Overall survival (OS) | Up to 30 months
  OS is defined as time from the start of treatment until the date of death due to any cause.
Number and percentage of AEs in patients receiving Ceralasertib and Durvalumab combination | Up to 30 months
  The safety and tolerability profile of Ceralasertib and Durvalumab combination will be evaluated using vital signs, laboratory data, electrocardiograms (ECGs), and adverse event data

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.Yes,indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home